CLINICAL TRIAL: NCT06181084
Title: A Pilot Study Comparing LY3410738 Capsule and Tablet Formulations and Effect of a Low-fat Meal and a Proton Pump Inhibitor on the Single-dose Pharmacokinetics of LY3410738 Tablets in Healthy Adult Subjects
Brief Title: A Study Comparing Different Formulations of LY3410738 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-IDH-21004; I9Y-OX-JDHE (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Formulation, food effect, proton pump inhibitor
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: Groups 1 and 2 have a randomized, 2-way crossover design and Groups 3 and 4 have a fixed-sequence design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Tablet versus Capsule (Experimental): Treatment A: LY3410738 capsule on Day 1 as a single oral dose in the morning following a fast of at least 10 hours prior to and 4 hours after dosing.
  Treatment B: LY3410738 tablet on Day 4 as a single oral dose in the morning 10 hours prior to and 4 hours after dosing.
  Interventions: Drug: LY3410738
- Group 2: Food Effect Comparison Group (Experimental): Treatment B: LY3410738 table on Day 1 as a single oral dose in the morning following a fast of at least 10 hours prior to and 4 hours after dosing.
  Treatment C: LY3410738 table on Day 4 as a single oral dose in the morning 30 minutes after starting a standard low-fat meal.
  Interventions: Drug: LY3410738
- Group 3: Potential of Hydrogen (pH) Effect Fasted Group (Experimental): Treatment B: LY3410738 table on Day 1 as a single oral dose in the morning following a fast of at least 10 hours prior to and 4 hours after dosing.
  Treatment D: Esomeprazole single oral dose once daily (QD) in the morning on Days 4 through 8 in fasted state followed by a standard low-fat meal. On Day 9, Esomeprazole a single oral dose followed by LY3410738 tablet as a single oral dose in the morning, following a fast of at least 10 hours prior to and 4 hours after esomeprazole and LY3410738 coadministration.
  Interventions: Drug: LY3410738; Drug: Esomeprazole
- Group 4: pH Effect Fed Group (Experimental): Treatment C: LY3410738 table on Day 1 as a single oral dose in the morning 30 minutes after starting a standard low-fat meal.
  Treatment E: Esomeprazole as a single oral dose QD in the morning on Days 4 through 8, in fasted state followed by a standard low-fat meal. On Day 9, Esomeprazole as a single oral dose followed by a LY3410738 tablet in the morning in fed state standard low-fat meal.
  Interventions: Drug: LY3410738; Drug: Esomeprazole

INTERVENTIONS:
Drug: LY3410738 — Administered orally.
Drug: Esomeprazole — Administered orally.
  Arms: Group 3: Potential of Hydrogen (pH) Effect Fasted Group; Group 4: pH Effect Fed Group

SUMMARY:
The main purpose of study is to compare different formulations of LY3410738 under fasting condition by looking at the amount of the study drug, LY3410738, that gets into the blood stream and how long it takes the body to get rid of it when given in healthy adult participants. The study will also access the effect of standard low-fat meal and esomeprazole (Proton Pump Inhibitor) on LY3410738. Safety and tolerability of LY3410738 will also be evaluated. For each participant, the total duration of the study will be 56 days for Groups 1 and 2 and up to 61 days for Groups 3 and 4, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m^2), inclusive.
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator.
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods.
* Must have comply with all study procedures, including the 3-night stay at the Clinical Research Unit (CRU) and follow-up phone call.

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor.
* Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B virus immunoglobulin M (HBV IgM) core antibody, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening.
* Positive polymerase chain reaction (PCR) test for COVID-19 at Screening.
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
* Have previously received LY3410738 in any other study investigating LY3410738, within 30 days prior to Day 1.
* Have history of a major surgical procedure within 30 days prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration-Time Curve from Hour 0 to the Last Measurable Concentration (AUC0-tlast) of LY3410738 Tablets Versus Capsules | Predose up to 48 hours postdose
  PK: AUC0-tlast of LY3410738 Tablets Versus Capsules
PK: Area Under the Concentration from Hour 0 Extrapolated to Infinity (AUC0-∞) of LY3410738 Tablets Versus Capsules | Predose up to 48 hours postdose
  PK: AUC0-∞ of LY3410738 Tablets Versus Capsules
PK: Maximum Observed Plasma Concentration (Cmax) of LY3410738 Tablets Versus Capsules | Predose up to 48 hours postdose
  PK: Cmax of LY3410738 Tablets Versus Capsules
PK: AUC0-tlast of LY3410738 After Standard Low-Fat Meal | Predose up to 48 hours postdose
  PK: AUC0-tlast of LY3410738 After Standard Low-Fat Meal
PK: AUC0-∞ of LY3410738 After Standard Low-Fat Meal | Predose up to 48 hours postdose
  PK: AUC0-∞ of LY3410738 After Standard Low-Fat Meal
PK: Cmax of LY3410738 After Standard Low-Fat Meal | Predose up to 48 hours postdose
  PK: Cmax of LY3410738 After Standard Low-Fat Meal
PK: AUC0-tlast of LY3410738 after Esomeprazole oral dose in the Fasted State | Predose up to 48 hours postdose
  PK: AUC0-tlast of LY3410738 after Esomeprazole oral dose in the Fasted State
PK: AUC0-∞ of LY3410738 after Esomeprazole oral dose in the Fasted State | Predose up to 48 hours postdose
  PK: AUC0-∞ of LY3410738 after Esomeprazole oral dose in the Fasted State
PK: Cmax of LY3410738 after Esomeprazole oral dose in the Fasted State | Predose up to 48 hours postdose
  PK: Cmax of LY3410738 after Esomeprazole oral dose in the Fasted State
PK: AUC0-tlast of LY3410738 after Esomeprazole oral dose in the Fed State | Predose up to 48 hours postdose
  PK: AUC0-tlast of LY3410738 after Esomeprazole oral dose in the Fed State
PK: AUC0-∞ of LY3410738 after Esomeprazole oral dose in the Fed State | Predose up to 48 hours postdose
  PK: AUC0-∞ of LY3410738 after Esomeprazole oral dose in the Fed State
PK: Cmax of LY3410738 after Esomeprazole oral dose in the Fed State | Predose up to 48 hours postdose
  PK: Cmax of LY3410738 after Esomeprazole oral dose in the Fed State

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, Study Director — Loxo Oncology, Inc.
Locations (1):
- Labcorp Clinical Research, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No